CLINICAL TRIAL: NCT02363634
Title: A Randomized Double Blind Parallel Group Placebo Controlled Clinical Trial Evaluating the Effects of Magtein on Anxiety, Mood and Sleep Quality in Older Adults
Brief Title: Clinical Trial to Evaluate Magtein in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miami Research Associates (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AIDP-Mg-2012
Record Dates: First submitted 2015-02-04; First posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Mood; Anxiety
Keywords: magnesium status; sleep quality
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — threonic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium threonate (Magtein) (Active Comparator): Those randomized to receive the Magtein
  Interventions: Dietary Supplement: magnesium threonate
- Placebo (Placebo Comparator): Those randomized to placebo

INTERVENTIONS:
Dietary Supplement: magnesium threonate — nutritional product
  Other Names: Magtein
  Arms: Magnesium threonate (Magtein)

SUMMARY:
A randomized double blind placebo controlled trial to evaluate the effects of a specialized magnesium on mood states and sleep quality in older adults.

DETAILED DESCRIPTION:
Efficacy Objectives:

To determine the effects of 12-weeks supplementation with Magtein™ as compared to placebo on:

1. anxiety and mood as measured by the Hamilton Anxiety Rating Scale (HAM-A) and the Positive and Negative Affect Schedule (PANAS). For the HAM-A, total score and sub-scores anxious mood, tension, fears, insomnia and intellectual will be utilized.
2. quality of sleep as measured by the Pittsburgh Sleep Quality Index (PSQI).
3. cognitive abilities as measured by the Erikson Flanker Task and computerized cognitive tests including Short-Term Memory Test (STM), Working Memory Test (WM), cued name recall task and face-name association task.

To determine the acute effects and the effects of 12-weeks supplementation with Magtein™ as compared to placebo on magnesium status as measured by the sponsor's protocol for determining body magnesium status.

Safety Objective:

To determine if supplementation with Magtein™ is safe within the confines of this study as denoted by changes from baseline to 12 weeks in blood work (comprehensive metabolic panel, uric acid and complete blood count with differential), blood pressure (BP), heart rate (HR), adverse events and subjective remarks.

ELIGIBILITY:
Inclusion Criteria

1. Subject is aged 45 to 70 years
2. Subject weighs between 50 and 100 kg.
3. Subject complains of having changes in their memory and concentration abilities.
4. Subject scores ≥ 12 and ≤ 28 on the Hamilton Anxiety Rating Scale (HAM-A)
5. Subject scores > 5 on the Pittsburgh Sleep Quality Index (PSQI)
6. Subject scores ≥ 24 on the Mini-Mental State Examination (MMSE) for the purpose of ruling out dementia and Alzheimer's disease
7. Female subject is surgically sterile, post-menopausal or agrees to use an acceptable method of birth control as defined in section 2.6.
8. Subject agrees to stop taking any vitamins, minerals, or dietary/herbal supplements he/she is currently taking at least 7 days prior to randomization and to not take any vitamins, minerals or dietary/herbal supplements other than the study product until after study completion.
9. Subject is willing and able to comply with the protocol including:

   * attending 4 visits, each of which are about 3 hours long;
   * not drinking alcohol or exercising for the 24 hours prior to the visits;
   * and not taking any vitamin, mineral, dietary or herbal supplements throughout the study.
10. Subject is able to understand and sign the informed consent to participate in the study.

Exclusion Criteria

1. Subject has any of the following medical conditions:

   * active heart disease
   * uncontrolled high blood pressure (≥ 140/90 mmHg)
   * renal or hepatic impairment/disease
   * Type I or II diabetes
   * bipolar disorder
   * Parkinson's disease
   * Alzheimer's disease
   * dementia
   * unstable thyroid disease
   * diagnosed major affective disorder
   * psychiatric disorder (hospitalized in the past year)
   * immune disorder (such as HIV/AIDS)
   * any medical condition deemed exclusionary by the Principal Investigator (PI)
2. Subject has a history of cancer (except localized skin cancer without metastases or in situ cervical cancer) within 5 years prior to screening.
3. Subject is currently taking calcium channel blockers, SSRI's or anxiolytics other than benzodiazepines as needed, with "as needed" defined as less than 5 times per month.
4. Subject is currently taking any medications that are known to interact with magnesium (see section 2.5.2).
5. Subject is currently taking antibiotics as the study product may reduce the absorption of antibiotics. A washout period of 2 weeks is allowed.
6. Subject is on an unstable dose of medication (defined as fewer than 90 days at the same dose).
7. Subject is currently taking any medication deemed exclusionary by PI.
8. Subject has an allergy or sensitivity to any ingredient in the test product (see section 3.2.1).
9. Subject exhibits evidence of hepatic or renal dysfunction as evidenced by ALT, AST, AP being ≥ 2 times the upper limit of normal or serum creatinine value ≥ 2.0 mg/dl or other clinically significant abnormal clinical laboratory value per PI discretion.
10. Subject has a history of drug or alcohol abuse in the past 12 months.
11. Subject has begun/stopped smoking ≤ 6 months ago OR has plans to begin/quit smoking.
12. Subject is pregnant, lactating, or planning to become pregnant during the study period.
13. Subject has any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the subject or the quality of the study data.
14. Subject is participating or has participated in another research study within 30 days prior to the screening visit

    -

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To determine the acute effects and the effects of 12-weeks supplementation with Magtein™ as compared to placebo on magnesium status as measured by the sponsor's protocol for determining body magnesium status. | 12 weeks
  To determine the acute effects and the effects of 12-weeks supplementation with Magtein™ as compared to placebo on magnesium status as measured by the sponsor's protocol for determining body magnesium status.

SECONDARY OUTCOMES:
To determine the effects of Magtein on Mood states ( as measured by the Hamilton Anxiety Rating Scale (HAM-A)) | 12 Weeks
  anxiety and mood as measured by the Hamilton Anxiety Rating Scale (HAM-A). For the HAM-A, total score and sub-scores anxious mood, tension, fears, insomnia and intellectual will be utilized.
To determine the effects of Magtein on Mood states ( As measured by the Positive and Negative Affect Schedule (PANAS) | 12 Weeks
  anxiety and mood as measured by the Positive and Negative Affect Schedule (PANAS).
To determine the effects of Magtein on sleep quality (as measured by the Pittsburgh Sleep Quality Index (PSQI) | 12 Weeks
  quality of sleep as measured by the Pittsburgh Sleep Quality Index (PSQI).
4. To determine the effects of Magtein on cognitive function (as measured by the Erikson Flanker Task) | 12 Weeks
  cognitive abilities as measured by the Erikson Flanker Task
4. To determine the effects of Magtein on cognitive function (as measured by computerized cognitive tests including Short-Term Memory Test (STM)) | 12 Weeks
  cognitive abilities as measured by computerized cognitive tests including Short-Term Memory Test (STM), Working Memory Test (WM), cued name recall task and face-name association task.
To determine relative safety of Magtein with 12 weeks use | 12 Weeks
  To determine if supplementation with Magtein™ is safe within the confines of this study as denoted by changes from baseline to 12 weeks in blood work (comprehensive metabolic panel, uric acid and complete blood count with differential), blood pressure (BP), heart rate (HR), adverse events and subjective remarks.

CONTACTS AND LOCATIONS:
Locations (1):
- Miami Research Associates, Miami, Florida, United States